CLINICAL TRIAL: NCT04877808
Title: Incidence and Predictive Value of Bacterial Surinfections on In-hospital Mortality in COVID-19 ICU Patients: a Longitudinal Single-center Study
Brief Title: Bacterial Surinfections in COVID-19 ICU Patients
Status: Completed | Type: Observational
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Principal Investigator, Jessa Hospital
Other Study IDs: f2021/037
Record Dates: First submitted 2021-05-03; First posted 2021-05-07 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to assess the incidence of bacterial surinfections (sepsis, VAP and catheter infections) in COVID-19 patients admitted to the ICU from 13th of March 2020 until 17h of October 2020. In addition, the association of these infections with the dose of corticosteroids, the length of stay in ICU and in hospital, the presence of venous thromboembolism, the number of bacterial episodes, the different types of bacteria causing the infections and ICU mortality will be evaluated as well as the associations between the presences of thrombi and bacteremia/catheter sepsis.

DETAILED DESCRIPTION:
Approximately 5% of patients with respiratory impairment develop a severe form with acute respiratory failure and require specialized management in the Intensive Care Unit (ICU). Invasive mechanical ventilation (IVM) exposes ICU patients to a particular risk of a nosocomial infectious complication called ventilator-associated pneumonia (VAP). In Europe, the incidence density is 18.3 VAP per 1000 days of IMV.

The coronavirus disease (COVID-19), caused by the severe acute respiratory syndrome coronavirus 2 (SARS CoV-2) emerged in December 2019 and has rapidly spread worldwide (Liu). The mortality of critical ill patients with COVID-19 has been reported variously as low as 11% and as high as 61% (Liu). Since March 2020, several thousand people have been receiving IMV due to severe COVID-19.

Informal exchanges between clinicians regarding the current pandemic indicate a high frequency of VAP. Several factors may account for a higher incidence of VAP in the population hospitalized in the ICU for SARS CoV-2 infection (Blonz 2021):

* A longer ventilation period, leading to greater mechanical exposure to the risk of VAP.
* The frequency of comorbidities.
* The frequency of ARDS, which is associated with a higher incidence of VAP.
* A form of acquired immunosuppression related to SARS-CoV-2 infection,
* Organizational factors related to the fact that this is the first major pandemic in modern history

Aim The aim of this study is to assess the incidence of bacterial surinfections (sepsis, VAP and catheter infections) in COVID-19 patients admitted to the ICU from 13th of March 2020 until 17h of October 2020. In addition, the association of these infections with the dose of corticosteroids, the length of stay in ICU and in hospital, the presence of venous thromboembolism, the number of bacterial episodes, the different types of bacteria causing the infections and ICU mortality will be evaluated as well as the associations between the presences of thrombi and bacteremia/catheter sepsis.

Design This is a retrospective, single-center study investigating the incidence of bacterial surinfections in COVID-19 patients admitted to the ICU from 13th of March 2020 until 17th of October 2020.

Inclusion criteria All adult COVID-19 patients admitted to the ICU from 13th of March until 17th of October 2020 were included.

Outcome measures The primary endpoint of this retrospective study is to assess the incidence of bacterial surinfections (sepsis, VAP and catheter infections) in COVID-19 patients admitted to the ICU from 13th of March 2020 until 17th of October 2020.

Secondary endpoints are the association of these infections with the dose of corticosteroids, the length of stay in ICU and in hospital, the presence of venous thromboembolism, the number of bacterial episodes, the different types of bacteria causing the infections and ICU mortality as well as the associations between the presences of thrombi and bacteremia/catheter sepsis in COVID-19 patients admitted to the ICU between 13th of March 2020 until 17th of October 2020.

Additional data collection

Additional collected parameters are listed below and are collected as a standard-of-care in our hospital:

* Demographics: i.e age, gender, BMI
* DNR code
* Comorbidities: smoking, obesity, hypertension, diabetes, cardiovascular disease, respiratory disease, malignancies, renal failure (AKI), liver failure, gastrointestinal disease, neurological conditions, mental state, other
* Symptoms at the time of admission to ICU: i.e fever, body temperature, dyspnoea, headache, diarrhea etc…
* Laboratory results of all standard parameters measured
* Treatment: antiviral agents, antibiotics, corticosteroids, etc…
* Complications: shock, heart failure, sepsis, stroke, bacteraemia, VAP, type of bacteria causing the infection, … etc
* Ventilation: method, PEEP, FiO2, P/F ratio ..
* Radiological findings: pneumonia, ground-glass opacity..

ELIGIBILITY:
Inclusion Criteria:

* All adult COVID-19 patients admitted to the ICU from 13th of March until 17th of October 2020 were included.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult COVID-19 patients admitted to the ICU from 13th of March until 17th of October 2020 were included.
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Incidence of sepsis | through study completion, 8 months
  Incidence of bacterial surinfections (sepsis) in COVID-19 patients admitted to the ICU
Incidence of VAP | through study completion, 8 months
  Incidence of bacterial surinfections (VAP) in COVID-19 patients admitted to the ICU
Incidence of bacterial catheter infections | through study completion, 8 months
  Incidence of bacterial surinfections (catheter infections) in COVID-19 patients admitted to the ICU

SECONDARY OUTCOMES:
Correlation with corticosteroids | through study completion, 8 months
  Correlation of bacterial surinfections with the dose of cortisosteroids
Correlation with the length of stay in ICU and hospital | through study completion, 8 months
  Correlation of bacterial surinfections with the length of stay in ICU and hospital
Correlation with venous thromboembolism | through study completion, 8 months
  Correlation of bacterial surinfections with the presence of venous thromboembolism
Correlation with the number of bacterial episodes | through study completion, 8 months
  Correlation of bacterial surinfections with the number of bacterial episodes
Correlation with the types | through study completion, 8 months
  Correlation with the different types of bacteria
Correlation with ICU mortality | through study completion, 8 months
  Correlation of bacterial surinfections with the ICU mortality
Correlation between presences of thrombi and bacteremia/catheter sepsis | through study completion, 8 months
  Correlation between presences of thrombi and bacteremia/catheter sepsis

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa hospital, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No
None sharing